CLINICAL TRIAL: NCT05882279
Title: Evaluation of the Effectiveness of Risk Minimization Measures: A Survey Among Pharmacists to Assess the Impact of the RMP Material for Patients on Promoting the Proper Use of NINLARO in Japan
Brief Title: A Survey on NINLARO Risk Management Plan (RMP) Material Utilization Among Pharmacists in Japan
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: C16065
Record Dates: First submitted 2023-05-22; First posted 2023-05-31 (Actual); Results first posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-05

CONDITIONS: Multiple Myeloma
Keywords: Drug Therapy
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pharmacists in Hospitals Prescribing NINLARO: Pharmacists included in Nikkei Research Access Panel who are active in clinical practice, with valid contact and who have instructed the dosing of NINLARO IRD therapy to patients with rrMM will self-administer a web-based survey. The questionnaires in the survey will be provided in Japanese.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
This is a survey among pharmacists who have instructed NINLARO therapy in ixazomib, lenalidomide and dexamethasone (IRD) dosing to patients with relapsed/refractory multiple myeloma (rrMM).

The main aims of the study are:

* To assess the frequency of pharmacists who have provided patients with the contents of the RMP material for patients.
* To assess the frequency of pharmacists who have obtained the RMP material for patients.
* To evaluate the depth of understanding of proper usage of NINLARO among pharmacists.

DETAILED DESCRIPTION:
This is a prospective, non-interventional, observational web-based survey in pharmacists who have instructed the dosing of NINLARO (ixazomib) in combination with lenalidomide and dexamethasone therapy to patients with rrMM. The study will assess the effectiveness of distributed RMP material in prevention of ixazomib overdose in Japanese clinical practice.

The study will enroll approximately 300 pharmacists who belong to hospitals prescribing NINLARO. The data will be collected through a self-administered web-based survey with questionnaires provided in Japanese.

This web-based survey will be conducted in Japan.

ELIGIBILITY:
Inclusion criteria:

1. Who belong to hospitals prescribing NINLARO.
2. Who have instructed the dosing of NINLARO in IRD therapy to patients.

Exclusion criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pharmacists included in Nikkei Research Access Panel, active in clinical practice, and with valid contact details who belong to hospitals prescribing NINLARO and instructed the dosing of NINLARO in IRD therapy to patients with rrMM will be randomly selected to participate in the survey.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/b6e2fa0988884fc1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment and response collection started on 01 June 2023 and ended on 09 June 2023.
Pre-assignment Details: A total of 24,000 pharmacists were requested to cooperate. Of these, 1329 pharmacists consented to participate in this study and 336 pharmacists passed the screening questions, out of which 6 pharmacists did not complete the questionnaire. 330 pharmacists were enrolled and completed all questions and were included in the analysis.
Groups:
- Pharmacists in Hospitals Prescribing NINLARO: Pharmacists included in Nikkei Medical Online Panel, active in clinical practice, and with valid contact details who belonged to hospitals and have instructed the dosing of NINLARO (ixazomib) in combination with lenalidomide and dexamethasone (IRD therapy) to patients were selected to participate in the survey.
Period: Overall Study
Arm/Group | Pharmacists in Hospitals Prescribing NINLARO
Started | 330
Completed | 330
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The final analysis set included all pharmacists who consented to participate in the survey, passed the screening questions, and completed all questions.
Arm/Group | Pharmacists in Hospitals Prescribing NINLARO
Number analyzed (Participants) | 330
Age, Customized [Count of Participants; unit: Participants] — Here, unit of measure: participants refer to pharmacists.
  Participants
    Greater than or equal to (>=) 22 years | 330
Sex: Female, Male [Count of Participants; unit: Participants] — Here, unit of measure: participants refer to pharmacists.
  Participants
    Female | 198
    Male | 132
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Here, unit of measure: participants refer to pharmacists.
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 330
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Here, unit of measure: participants refer to pharmacists.
  Participants
    American Indian or Alaska Native | 0
    Asian | 330
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 0
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants] — Here, unit of measure: participants refer to pharmacists.
  Participants
    Japan | 330

OUTCOME MEASURES:

1. Primary Outcome: Number of Pharmacists Who Had Provided Patients With the Contents of the Risk Management Plan (RMP) Material
Description: The NINLARO additional risk minimization measure (aRMM) effectiveness study questionnaire which was intended for pharmacists who instructed the dosing of IRD therapy to patients with relapsed/refractory multiple myeloma (RRMM). This outcome was based on the number of pharmacists who answered "Yes" to question 3; Do you instruct patients that they should take one capsule of NINLARO each time on an empty stomach for RRMM? Here, unit of measure: participants refer to pharmacists.
Time Frame: Up to Day 9
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacists in Hospitals Prescribing NINLARO
Number analyzed (Participants) | 330
Participants | 307

2. Secondary Outcome: Number of Pharmacists Who Had Received the RMP Material for Patients
Description: The NINLARO aRMM effectiveness study questionnaire which was intended for pharmacists who instructed the dosing of IRD therapy to patients with RRMM. This outcome was based on the number of pharmacists who answered "Yes" to question 7; Have you obtained the RMP material for patients? Here, unit of measure: participants refer to pharmacists.
Time Frame: Up to Day 9
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacists in Hospitals Prescribing NINLARO
Number analyzed (Participants) | 330
Participants | 124

3. Secondary Outcome: Number of Pharmacist With Understanding of the Proper NINLARO Dosing Schedule
Description: The NINLARO aRMM effectiveness study questionnaire which was intended for pharmacists who instructed the dosing of IRD therapy to patients with RRMM. This outcome was based on the number of pharmacists who answered "Yes" to question 1; Do you know that patients will take one capsule of NINLARO each time on an empty stomach for RRMM? Here, unit of measure: participants refer to pharmacists.
Time Frame: Up to Day 9
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacists in Hospitals Prescribing NINLARO
Number analyzed (Participants) | 330
Participants | 316

4. Secondary Outcome: Number of Pharmacist With Understanding of the Importance of Providing NINLARO Dosing Schedule
Description: The NINLARO aRMM effectiveness study questionnaire which was intended for pharmacists who instructed the dosing of IRD therapy to patients with RRMM. This outcome was based on question 2; Do you think it is important to inform patients that they should take one capsule of NINLARO each time on an empty stomach for RRMM? Here, unit of measure: participants refer to pharmacists.
Time Frame: Up to Day 9
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacists in Hospitals Prescribing NINLARO
Number analyzed (Participants) | 330
Participants
  Very important | 298
  Rather important | 30
  Rather not important | 1
  Not important | 1

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events data were not collected/assessed in this study
Description: This was a web-based multiple choice questionnaire survey of pharmacists which did not include safety information as adverse events were not planned to be collected in this study. Data '0' for total number of participants at risk/affected for sections all-cause mortality, serious adverse events, and other (not including serious adverse events) signifies that adverse events were not collected and assessed in this study.
Arm/Group | Pharmacists in Hospitals Prescribing NINLARO
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT05882279/Prot_SAP_000.pdf